CLINICAL TRIAL: NCT05012956
Title: Measuring Abdominal Wall Compliance During Gynecologic Laparoscopic Surgery
Acronym: AbComp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Jan Deprest, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S65329
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: Group 1: pelvic organ prolapse patients
  Group 2: patients assigned to gynecologic laparoscopic surgery, other than pelvic organ prolapse, at UZ Leuven.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POP group (Active Comparator): Pelvic organ prolapse patients enrolled for sacrocolpopexy surgery at UZ Leuven.
  Interventions: Procedure: Laparoscopic sacrocolpopexy
- Control group (Active Comparator): Patients assigned to gynecologic laparoscopic surgery, other than sacrocolpopexy, at UZ Leuven.
  Interventions: Procedure: gynecologic laparoscopic surgery

INTERVENTIONS:
Procedure: Laparoscopic sacrocolpopexy — During laparoscopic sacrocolpopexy, the anatomical position of the vaginal vault and cervix (if present) is restored by suturing a surgical mesh to the vaginal cuff or cervix and variable portions of the anterior and posterior vagina, while connecting the other end of the mesh to the anterior longitudinal ligament over the sacrum.
  Arms: POP group
Procedure: gynecologic laparoscopic surgery — Gynecologic laparoscopic surgery at UZ Leuven, other than sacrocolpopexy
  Arms: Control group

SUMMARY:
To measure abdominal wall compliance (AWC) during gynaecologic laparoscopy and assess its relation to the pelvic organ prolapse quantification (POP-Q) score of the same individual, and determine a relationship if present.

DETAILED DESCRIPTION:
To characterize abdominal wall compliance (AWC), sterile reflective markers are attached to the abdominal wall by means of surgical tape, and the movement of these markers will be tracked with an optical tracker device. As during normal surgery, the intra-abdominal pressure (IAP) measured by the insufflator device will be recorded and stored on a secure computer with dedicated software. The pelvic organ quantification (POP-Q) score for each patient is determined pre-surgery as part of the standard of care. A biomechanical model will use reflective marker displacement (RMD) and IAP to calculate AWC. The POP-Q score will then be used to investigate a relation between AWC and degree of prolapse.

It is important to state that the trial does not intervene with the standard of care before- and during surgery. The used equipment is non-invasive and only requires about 5 minutes to be set up before the start of surgery. This set up comprises placing the optical tracker in the operating room such that it has a line of sight on the patient's abdomen and attaching the sterile markers to the abdominal wall. Therefore the trail does not add any additional risk to the surgery.

Each patient scheduled for gynecologic laparoscopy will be asked to participate in the study. If the patient wants to participate, she is presented the informed consent form (ICF). If both patient and clinician in charge sign the ICF, the patient is included in the study. The table below shows the patient specific information stored as part of the study.

Sample size calculation is based on a previous study (S61346), where we measured vaginal wall stiffness (the inverse of compliance) in patients with varying degrees of prolapse. 20 POP patients and 20 control group patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* All patients assigned to gynecologic laparoscopic surgery at UZ Leuven.

Exclusion Criteria:

* Patients that are unable to give consent: In case of dementia or other cognitive disorders.
* Patients that are unable to give consent: When they are unable to read and/or interpret the content of the informed consent form (ICF), which is written in Dutch.
* Patients that had had an earlier abdominoplasty or abdominal wall mesh implantation, or other operations that directly affect the biomechanical properties of the abdominal wall.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Intra-abdominal pressure (IAC) | During surgery
  Measured as part of the surgery by the insufflator device. [mmHg]
Reflective marker displacement (RMD) | Druign surgery
  Measured by an infrared camera and reflective markers attached to the abdominal wall. [mm]

SECONDARY OUTCOMES:
Pelvic organ quantification score | pre-surgery examination
  Pelvic organ quantification (POP-Q) score, indicating the degree of pelvic organ prolapse (standardized method). The POP-Q score ranges from 0 (no prolapse) to IV (high prolapse). It is expected that a higher POP-Q score results in a higher abdominal wall compliance.
Age | pre-srugery
  Age of the patient
BMI | pre-surgery
  Body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- Ann-Sophie Page, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No